CLINICAL TRIAL: NCT00744679
Title: An Assessment of the Steady-State Pharmacokinetic and Pharmacodynamic Profile of Tysabri 300 mg Following at Least 12 Monthly Infusions
Brief Title: A Pharmacokinetic (PK) Study of Natalizumab (Tysabri) at Steady State
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 101MS406
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
Keywords: MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab 300 mg (Experimental): Natalizumab infused at 300 mg every 28 days during the screening and assessment periods of the study which continues the therapy of the previous 12 months and maintains steady-state pharmacokinetics.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Participants continue to receive regularly-scheduled doses of Tysabri (300 mg infusion every 28±7 days) through the Tysabri Outreach: United Commitment to Health Prescribing Program (TOUCH) throughout the screening and assessment periods. Participants must continue to be dosed every 28±7 days in order to maintain steady-state pharmacokinetics.
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective is to assess the pharmacokinetic (PK) profile of natalizumab (Tysabri) at steady state.

The secondary objective is to assess the pharmacodynamics (PD) profile (α4 integrin saturation) of Tysabri at steady state.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Must be a multiple sclerosis (MS) patient enrolled in the Tysabri Outreach: United Commitment to Health Prescribing Program (TOUCH) who is not expected to discontinue Tysabri therapy prior to completion of the requirements of this study.
* Must have been treated with monthly IV infusions of Tysabri 300 mg for at least 12 months, with the 9 most recent doses having been administered at 28±7 day intervals.
* Must test negative for antibodies to Tysabri at the Screening Visit.
* Must have a magnetic resonance imaging (MRI) brain scan, performed prior to the initiation of treatment with Tysabri, on file.
* Must weigh between 42 and 126 kg, inclusive.
* All male subjects and female subjects of childbearing potential must practice effective contraception during the study.

Key Exclusion Criteria:

* History of, or abnormal laboratory results indicative of, any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* Positive result for antibodies to Tysabri at any prior evaluation.
* Treatment with an investigational product or approved therapy for investigational use within 6 months prior to the start of PK sample collection or during the course of this study. Concurrent participation in an observational study (e.g., Tysabri Global Observational Program in Safety [TYGRIS]) is permitted.
* Pre-scheduled for any elective procedure or medical treatment during the study period.
* History of drug or alcohol abuse (as defined by the Investigator) within 2 years prior to the Screening Visit.
* Female subjects who are breastfeeding, pregnant, or planning to become pregnant while on study.
* Alcohol use within 24 hours prior to the Baseline Visit.
* Inability or unwillingness to comply with study requirements, including the presence of any condition (e.g., physical, mental, social) that is likely to affect the subject's ability to comply with the study protocol.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Profile of Natalizumab | Baseline (Day 0), 2 hours after infusion starts on Days 1 and on Days 2, 3, 4, 7, 14, 21 and 28

SECONDARY OUTCOMES:
Natalizumab Binding Saturation Of α4 Integrin Sites On Peripheral Blood Mononuclear Cells (PBMC). | Baseline (Day 0), 2 Hours after infusion starts on Days 1, and on Days 4, 7, 14, 21 and 28
  The pharmacodynamic activity of natalizumab is assessed by measuring the degree of natalizumab saturation of the VLA-4 (α4β1 integrin) receptor on peripheral blood lymphocyte/monocyte populations.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Latham, New York, United States